CLINICAL TRIAL: NCT01187381
Title: Multicenter, Single-Arm, Observational Study of Mean Duration of Trastuzumab (Herceptin) Treatment in Patients With HER2-Positive Early or Metastatic Breast Cancer in Romanian Population
Brief Title: An Observational Study of the Mean Duration of Trastuzumab (Herceptin) Treatment in Participants With Early or Metastatic Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Breast Cancer
Acronym: HERODOT
Status: Terminated | Type: Observational
Why Stopped: Study was prematurely terminated because of missing data collection.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25235
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Breast Cancer: Participants with early or metastatic HER2-positive breast cancer who were receiving treatment with trastuzumab according to local standard of care and in line with the current summary of product characteristics/ local guidelines, will be observed. Dosing and treatment duration of the trastuzumab will be at the discretion of the treating physician.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab according to local standard of care and in line with the current summary of product characteristics/ local guidelines
  Other Names: Herceptin

SUMMARY:
This single arm observational study will assess the duration and safety of treatment with trastuzumab in routine clinical practice in participants with early or metastatic HER2-positive breast cancer. Data will be collected from female participants treated with trastuzumab according to the Summary of Product Characteristics and local protocols. Duration of observation for each participant is from therapy initiation until permanent discontinuation for any cause.

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive breast cancer
* Treated with trastuzumab in accordance with Summary of Product Characteristics and local protocols
* Written informed consent to data collection

Exclusion Criteria:

* Any contraindication to trastuzumab
* Clinically relevant cardiovascular disorder or disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female participants with early or metastatic HER2-positive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-04-14 (Actual); Primary Completion 2015-10-15 (Actual); Study Completion 2015-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Cluj Clinical County Hospital; Oncology Dept, Cluj-Napoca, Romania

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Breast Cancer: Participants with early or metastatic human epidermal growth factor receptor 2 (HER2)-positive breast cancer who were receiving treatment with trastuzumab according to local standard of care and in line with the current summary of product characteristics/ local guidelines, were observed (overall observation period: 5 years). Dosing and treatment duration of the trastuzumab were at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Participants With Breast Cancer
Started | 250
Completed | 250 (A participant completed study when the trastuzumab treatment was discontinued.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Participants With Breast Cancer: Participants with early or metastatic HER2-positive breast cancer who were receiving treatment with trastuzumab according to local standard of care and in line with the current summary of product characteristics/ local guidelines, were observed (overall observation period: 5 years). Dosing and treatment duration of the trastuzumab were at the discretion of the treating physician.
Arm/Group | Participants With Breast Cancer
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2600 (10.61939)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Duration With Trastuzumab in the Routine Clinical Practice
Time Frame: Baseline up to 5 years
Population: Number of participant analyzed=participants with data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Participants With Breast Cancer
Number analyzed (Participants) | 246
Days | 401.90 (229.867)

2. Secondary Outcome: Percentage of Participants Who Discontinued Trastuzumab Therapy According to Reasons for Discontinuation
Time Frame: Baseline up to 5 years
Population: All enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Breast Cancer
Number analyzed (Participants) | 250
percentage of participants
  Adverse event | 5
  Death | 2
  Progression of the disease | 18
  Administrative reasons | 30
  Doctor's decision | 40
  Other Than the Reasons Reported Above | 5

3. Secondary Outcome: Percentage of Participants Who Received Previous Neoadjuvant Therapy
Description: As a neoadjuvant therapy, participants received chemotherapy alone, radiotherapy alone, hormonal therapy alone or combination of these therapies. Percentage of participants who received these therapies is reported.
Time Frame: Baseline up to 5 years
Population: Number of participants analyzed=participant with data available for this outcome
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Breast Cancer
Number analyzed (Participants) | 210
percentage of participants
  Chemotherapy and Radiotherapy | 28
  Chemotherapy and Radiotherapy and Hormonal therapy | 28
  Chemotherapy and Hormonal therapy | 8
  Radiotherapy and Hormonal therapy | 7
  Chemotherapy alone | 21
  Radiotherapy alone | 6
  Hormonal therapy alone | 2

4. Secondary Outcome: Percentage of Participants Who Had Surgical Procedure for Breast Cancer
Description: Percentage of participants who underwent different types of surgical procedures for breast cancer are reported. Different types of surgical procedures included: breast-conserving surgery; mastectomy; and other (any other surgical procedure except breast-conserving surgery and mastectomy).
Time Frame: Baseline up to 5 years
Population: Number of participants analyzed=participants who were evaluable for this outcome measure
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Breast Cancer
Number analyzed (Participants) | 237
percentage of participants
  Breast-conserving surgery | 21.2
  Mastectomy | 73.2
  Other | 0.4

5. Secondary Outcome: Percentage of Participants Who Received Trastuzumab as Adjuvant Therapy of HER2 Positive Breast Cancer
Time Frame: Baseline up to 5 years
Population: All enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Breast Cancer
Number analyzed (Participants) | 250
percentage of participants | 82

6. Secondary Outcome: Progression Free Survival
Description: Progression free survival was defined as the time from first dose of trastuzumab to disease progression as assessed by treating physician. Due to observational nature of the study, there was no specific method of assessment used to define progressive disease. Progressive disease was confirmed by treating physician, based on his/her assessment according to local practice.
Time Frame: Baseline uo tp 5 years
Population: Number of participants analyzed=participants who presented progression of disease
Measure: Median (Full Range); unit: days
Arm/Group | Participants With Breast Cancer
Number analyzed (Participants) | 44
days | 324 [84 to 1849]

7. Secondary Outcome: Percentage of Participants by the Site of First Disease Progression
Time Frame: Baseline up to 5 years
Population: Number of participants analyzed=participants who presented disease progression
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Breast Cancer
Number analyzed (Participants) | 44
percentage of participants
  Bone | 11
  Brain | 32
  Breast | 9
  Liver | 27
  Lung | 21

ADVERSE EVENTS:
Time Frame: Baseline up to 5 years
Arm/Group | Participants With Breast Cancer
Serious Adverse Events (participants affected / at risk) | 12/250
Other Adverse Events (participants affected / at risk) | 17/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Breast Cancer (N=250)
Cardiac failure chronic (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Chills (General disorders) | 1
Death (General disorders) | 1
Metastases to liver (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Hepatitis viral (Hepatobiliary disorders) | 1
Ejection fraction decreased (Investigations) | 2
Craniofacial fracture (Musculoskeletal and connective tissue disorders) | 1
Transient ischemic attack (Nervous system disorders) | 1
Breast cancer metastatic (Reproductive system and breast disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Breast Cancer (N=250)
Leukopenia (Blood and lymphatic system disorders) | 2
Edema peripheral (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 2
Ejection fraction decreased (Investigations) | 4
Craniofacial fracture (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Herpes zoster (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Study was prematurely terminated because of missing data collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.